CLINICAL TRIAL: NCT02901977
Title: On the Antithrombotic Effects of Doxazosin and Ramipril in Essential Hypertension
Brief Title: Doxazosin and Ramipril in Hypertension
Acronym: DoRa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Thomas Kahan, Principal investigator, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-000631-25
Record Dates: First submitted 2016-09-09; First posted 2016-09-15 (Estimated); Last update posted 2025-03-04 (Actual); Status verified 2016-09

CONDITIONS: Hypertension
Keywords: Hypertension; Blood pressure; Hemostasis; Endothelial function
MeSH Terms: conditions — Hypertension | interventions — Ramipril; Doxazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACE inhibitor (Experimental): Ramipril tablets 10 mg od for 12 weeks
  Interventions: Drug: Ramipril
- Alpha receptor blocker (Active Comparator): Doxazosin tablets 8 mg od for 12 weeks
  Interventions: Drug: Doxazosin

INTERVENTIONS:
Drug: Ramipril — Antihypertensive therapy
  Other Names: Tiratec
  Arms: ACE inhibitor
Drug: Doxazosin — Antihypertensive therapy
  Other Names: Alfadil ,Cardura
  Arms: Alpha receptor blocker

SUMMARY:
Randomized double-blind parallel group study in patients with mild-to-moderate hypertension to evaluate the effects beyond the blood pressure lowering effect of treatment for 12 weeks with ramipril or doxazosin on hemostatic mechanisms and on endothelial function.

DETAILED DESCRIPTION:
This study aims to answer the following questions: 1) Does antihypertensive therapy with doxazosin exhibit antithrombotic effects in patients with essential hypertension? 2) Are the potential antithrombotic effects of doxazosin different to the effects of an ACE inhibitor? 3) Is there a relation between the antihypertensive effect and the antithrombotic effect of these antihypertensive agents?

The co-primary outcomes are changes in endothelial function assessed by flow mediated vasodilatation, and in haemostatic function measured by the generation of thrombin-antithrombin complex.

ELIGIBILITY:
Inclusion Criteria:

* Primary mild-to-moderate hypertension

Exclusion Criteria:

* Pregnancy and lactation
* Recent (6 months) malignant disease or ongoing treatment for malignancy
* No absolute indication or contraindication for any of the study drugs

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-03; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Thrombin generation | 12 weeks
  Thrombin-Antithrombin complex (TAT)
Endothelial function | 12 weeks
  Forearm post-ischemic flow mediated dilatation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kahan, MD, Principal Investigator — Karolinska Institutet, Department of Clinical Sciences, Danderyd Hospital
Locations (1):
- Karolinska Institutet, Daprtment of Clinical Sciences, Danderyd Hospital, Cardiovascular Research Laboratory, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jekell A, Kalani M, Kahan T. The interrelation of endothelial function and microvascular reactivity in different vascular beds, and risk assessment in hypertension: results from the Doxazosin-ramipril study. Heart Vessels. 2019 Mar;34(3):484-495. doi: 10.1007/s00380-018-1265-7. Epub 2018 Sep 22. PMID 30244381
- [Derived] Ekholm M, Jekell A, Wallen NH, Gigante B, Kahan T. Effects of Angiotensin-Converting Enzyme Inhibition and Alpha 1-Adrenergic Receptor Blockade on Inflammation and Hemostasis in Human Hypertension. J Cardiovasc Pharmacol. 2018 Apr;71(4):240-247. doi: 10.1097/FJC.0000000000000565. PMID 29389738
- [Derived] Jekell A, Kahan T. The usefulness of a single arm cuff oscillometric method (Arteriograph) to assess changes in central aortic blood pressure and arterial stiffness by antihypertensive treatment: results from the Doxazosin-Ramipril Study. Blood Press. 2018 Apr;27(2):88-98. doi: 10.1080/08037051.2017.1394791. Epub 2017 Oct 26. PMID 29073803
- [Derived] Jekell A, Kalani M, Kahan T. The effects of alpha 1-adrenoceptor blockade and angiotensin converting enzyme inhibition on central and brachial blood pressure and vascular reactivity: the doxazosin-ramipril study. Heart Vessels. 2017 Jun;32(6):674-684. doi: 10.1007/s00380-016-0924-9. Epub 2016 Nov 24. PMID 27885499